CLINICAL TRIAL: NCT00470158
Title: Delivery of Iron and Zinc Supplements: Evaluation of Interaction Effect on Biochemical and Clinical Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H.22.05.03.11.C2; GHS-A-00-03-00019-00-90027844
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2011-09-19 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2009-12

CONDITIONS: Anemia; Diarrhea; Iron
Keywords: zinc; iron; interaction; diarrhea; delivery
MeSH Terms: conditions — Anemia; Diarrhea | interventions — Iron; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- combined iron and zinc (Experimental): Iron and zinc together
  Interventions: Dietary Supplement: iron and zinc combined
- Separate iron and zinc (Experimental): Iron and zinc on separate days
  Interventions: Dietary Supplement: iron and zinc on separate days
- iron alone (Experimental): Iron
  Interventions: Dietary Supplement: iron
- zinc alone (Experimental): Zinc
  Interventions: Dietary Supplement: Zinc
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: iron and zinc combined — Children >= 12 months received an average of 5mg zinc/day, 6.25 Iron/day, and 25IU folic acid/day. children<12 received half that dose. This dose was alternated daily with placebo. Dissolvable doses were distributed in blister packs and reconstituted with a teaspoon of water. Doses were administered in the morning. For missed doses, the mother gave the child the next morning dose, and a second dose in the evening.
  Other Names: Tablets were manufactured by Nutriset; S.A.S. (Malaunay, France).
  Arms: combined iron and zinc
Dietary Supplement: iron and zinc on separate days — Children >= 12 months received an average of 5mg zinc/day, alternating daily with 6.25 Iron/day, and 25IU folic acid/day. Children<12 received half that dose. Dissolvable doses were distributed in blister packs and reconstituted with a teaspoon of water. Doses were administered in the morning. For missed doses, the mother gave the child the next morning dose, and a second dose in the evening.
  Other Names: Tablets were manufactured by Nutriset; S.A.S. (Malaunay, France).
  Arms: Separate iron and zinc
Dietary Supplement: iron — Children >= 12 months received an average 6.25 Iron/day, and 25IU folic acid/day. Children<12 received half that dose. This dose was alternated daily with placebo. Dissolvable doses were distributed in blister packs and reconstituted with a teaspoon of water. Doses were administered in the morning. For missed doses, the mother gave the child the next morning dose, and a second dose in the evening.
  Arms: iron alone
Dietary Supplement: Zinc — Children >= 12 months received an average of 5mg zinc/day. Children<12 received half that dose. This dose was alternated daily with placebo. Dissolvable doses were distributed in blister packs and reconstituted with a teaspoon of water. Doses were administered in the morning. For missed doses, the mother gave the child the next morning dose, and a second dose in the evening.
  Arms: zinc alone
Dietary Supplement: placebo — Children received daily placebo. Dissolvable doses were distributed in blister packs and reconstituted with a teaspoon of water. Doses were administered in the morning. For missed doses, the mother gave the child the next morning dose, and a second dose in the evening.
  Arms: placebo

SUMMARY:
With the long-term public health goal of developing an effective micronutrient supplementation program to improve child health by improving iron and zinc status and decreasing morbidity due to diarrhea in areas with high rates of childhood malnutrition, we seek to determine the most efficacious method of decreasing childhood morbidity and mortality due to diarrhea in toddlers by re-examining the issue of iron and zinc interaction and determining if this interaction can be minimized by separate administration of iron and zinc supplementation.

DETAILED DESCRIPTION:
Iron supplementation is used in reducing anemia and improving hemoglobin status. Zinc supplementation is emerging as possibly an efficacious preventive measure in decreasing incidence of severe diarrhea. Previous studies have suggested interactions of zinc and iron when given together, reducing the effects of supplementation with both minerals. One study in Peru has shown a decrease in interaction effect with separate supplementation of iron and zinc in time when compared to iron administration alone or placebo; however, an evaluation of clinical outcomes and zinc or iron status when iron and zinc are administered separately compared to supplementation of zinc and iron together or each alone has not previously been done. This trial will assess the effect of iron and zinc supplementation given on alternate days compared with giving them together in a combined supplement.

We propose a randomized, double blind, placebo-controlled community trial of children 6-23 months in Mirzapur, Bangladesh. We will recruit and enroll 1000 children 6-23 months old who are permanent residents of the selected villages. Each child will be randomly assigned to 1) daily alternating zinc and placebo 2) daily alternating iron/folic acid and placebo 3) daily alternating zinc/iron/folic acid and placebo 4) daily alternating zinc and iron/folic acid 5) daily placebo. Primary outcomes will include incidence of severe diarrhea, evaluated weekly for 6 months, hemoglobin, prevalence of anemia, and serum zinc.

Analysis of the data will be done to compare the effect of separate iron and zinc supplementation as compared to combined iron and zinc supplementation as well as compared to iron, zinc, or placebo single supplementation. We will evaluate the difference in incidence rate of severe diarrhea, serum hemoglobin, percent anemia, and serum zinc. Since this will be a randomized, double-blind, placebo controlled trial, differences in effect will be most likely explained by the timing of supplement doses. If there is an improvement in clinical and biochemical outcomes, this would be consistent with a decreased interaction of absorption. If no difference is found, there may be another mechanism for the seeming interaction of iron and zinc besides that of mutually inhibitory absorption in the intestine.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-18 months old
* Permanent residents of the selected villages

Exclusion Criteria:

* Severe malnutrition requiring hospitalization (defined as weight for height <-3 SD Z-score)
* Severe anemia requiring treatment (hemoglobin < 70 g/L)
* Chronic illness that would impair feeding ability
* Likely to move in next 6 months.
* Fever greater than 38.5
* Regular iron supplementation

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Black, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- ICDDR,B, Dhaka, Mohakhali, Bangladesh

REFERENCES:
- [Result] Chang S, El Arifeen S, Bari S, Wahed MA, Rahman KM, Rahman MT, Mahmud AB, Begum N, Zaman K, Baqui AH, Black RE. Supplementing iron and zinc: double blind, randomized evaluation of separate or combined delivery. Eur J Clin Nutr. 2010 Feb;64(2):153-60. doi: 10.1038/ejcn.2009.127. Epub 2009 Nov 11. PMID 19904293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 6-18 month old permanent residents of selected villages near Kumudini Hospital were enrolled from May 8, 2007-August 31, 2007.
Pre-assignment Details: If one family had two eligible children, one was randomly selected for enrollment. Children with severe malnutrition (weight for height z-score -3 s.d.), severe anemia (hemoglobin <70 g/l), chronic illnesses that would impair feeding ability, planned move during the study period, or active fever (>38.5 C) were excluded from the study.
Groups:
- Combined Iron and Zinc: combined iron and zinc, alternating daily with placebo
- Separate Iron and Zinc: iron, alternating daily with zinc
- Iron Alone: iron, alternating daily with placebo
- Zinc Alone: zinc, alternating daily with placebo
- Placebo: placebo daily
Period: Overall Study
Arm/Group | Combined Iron and Zinc | Separate Iron and Zinc | Iron Alone | Zinc Alone | Placebo
Started | 201 (9 children received wrong samples at enrollment and were analyzed by the supplement received.) | 199 (9 children received wrong samples at enrollment and were analyzed by the supplement received.) | 201 (9 children received wrong samples at enrollment and were analyzed by the supplement received.) | 198 (9 children received wrong samples at enrollment and were analyzed by the supplement received.) | 201 (9 children received wrong samples at enrollment and were analyzed by the supplement received.)
Completed | 193 (Enrolled for at least 90% of total study time.) | 191 (Enrolled for at least 90% of total study time.) | 193 (Enrolled for at least 90% of total study time.) | 193 (Enrolled for at least 90% of total study time.) | 195 (Enrolled for at least 90% of total study time.)
Not Completed | 8 | 8 | 8 | 5 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 7 | 8 | 8 | 5 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Iron and Zinc | Separate Iron and Zinc | Iron Alone | Zinc Alone | Placebo | Total
Number analyzed (Participants) | 201 | 199 | 201 | 198 | 201 | 1000
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 201 | 199 | 201 | 198 | 201 | 1000
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.93 (0.31) | 0.925 (0.32) | 0.9 (0.33) | 0.925 (0.33) | 0.9 (0.32) | 0.92 (0.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 107 | 93 | 109 | 88 | 484
  Male | 114 | 92 | 108 | 89 | 113 | 516
Region of Enrollment [Number; unit: participants]
  Bangladesh | 201 | 199 | 201 | 198 | 201 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Diarrhea
Description: A diarrhea episode was defined as three or more loose, liquid, or watery stools for 2 consecutive days, separated in time from an earlier or subsequent episode by at least 2 consecutive diarrhea-free days.
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Combined Iron and Zinc | Separate Iron and Zinc | Iron Alone | Zinc Alone | Placebo
Number analyzed (Participants) | 201 | 199 | 201 | 198 | 201
episodes | 201 | 204 | 260 | 224 | 235

2. Secondary Outcome: Change in Hemoglobin
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Zinc Status
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Percent Anemic
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Combined Iron and Zinc | Separate Iron and Zinc | Iron Alone | Zinc Alone | Placebo
Serious Adverse Events (participants affected / at risk) | 11/201 | 8/199 | 17/201 | 10/198 | 22/201
Other Adverse Events (participants affected / at risk) | 2/201 | 2/199 | 0/201 | 4/198 | 4/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Iron and Zinc (N=201) | Separate Iron and Zinc (N=199) | Iron Alone (N=201) | Zinc Alone (N=198) | Placebo (N=201)
infectious hospitalizations (Infections and infestations) | 11 | 8 | 17 | 10 | 22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Iron and Zinc (N=201) | Separate Iron and Zinc (N=199) | Iron Alone (N=201) | Zinc Alone (N=198) | Placebo (N=201)
noninfectious hospitalizations (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 0 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No